CLINICAL TRIAL: NCT07253948
Title: Distribution Characteristics of Helicobacter Pylori in Different Gastritis and Early Gastric Cancer States Using Immunohistochemical Staining
Brief Title: Distribution Characteristics of Helicobacter Pylori
Status: Recruiting | Type: Observational
Sponsor: Jilin University (Other)
Responsible Party: Principal Investigator, Dong Yang, Principal Investigator, Jilin University
Other Study IDs: 130029
Record Dates: First submitted 2025-11-13; First posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Helicobacter Pylori; Early Gastric Cancer
Keywords: Helicobacter pylori; Immunohistochemical staining; Atrophic gastritis; Early gastric cancer screening
MeSH Terms: conditions — Stomach Neoplasms; Gastritis, Atrophic

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- received H. pylori immunohistochemical testing at our center and tested positive
  Interventions: Diagnostic Test: immunohistochemical testing

INTERVENTIONS:
Diagnostic Test: immunohistochemical testing — Immunohistochemical results were reviewed independently by two experienced pathologists, with disagreements resolved by a third. Immunohistochemical staining was performed using an anti-H. pylori antibody (Beijing Zhongshan Golden Bridge Biotechnology Co., Ltd, Beijing, China). Positive results were graded as mild (1+): occasional bacteria or colonization in <1/3 of the specimen length; moderate (2+): colonization exceeding 1/3 but <2/3 of the specimen, or continuous but sparse distribution on the epithelial surface; and severe (3+): clusters of H. pylori distributed across the full length of the specimen. The gastric body and antrum were assessed separately, and distribution patterns were classified as gastric antrum > gastric body, gastric antrum = gastric body, or gastric body > gastric antrum. The distribution of H. pylori across subgroups was compared, and multivariate analyses were performed to identify risk factors associated with the development of early gastric cancer.

SUMMARY:
This study aimed to analyze the distribution characteristics of Helicobacter pylori（H. pylori） in varying stages of atrophic gastritis and early gastric cancer using immunohistochemical staining, with the goal of providing guidance for the early screening of gastric cancer.

A retrospective analysis was conducted on gastric biopsy cases that underwent H. pylori immunohistochemical staining at our center from March 1, 2023, to August 15, 2025. Cases were classified into non-atrophic and atrophic groups based on the presence or absence of gastric atrophy. All cases were further divided into non-open and open atrophy groups and additionally into early gastric cancer and non-cancer groups. The distribution of H. pylori across subgroups was compared, and multivariate analyses were performed to identify risk factors associated with the development of early gastric cancer.

DETAILED DESCRIPTION:
A retrospective analysis was performed on cases that underwent gastric H. pylori immunohistochemical staining at our center from March 1, 2023, to August 15, 2025.

Immunohistochemical results were reviewed independently by two experienced pathologists, with disagreements resolved by a third. After applying inclusion and exclusion criteria, cases were classified according to the Kimura-Takemoto classification : First, patients were categorized into non-atrophic and atrophic groups based on the presence of atrophy. Second, all cases were further divided into non-open and open atrophy groups. Open atrophy was defined as a degree of O1 or greater (endoscopic atrophic border extending beyond the cardia). All cases were additionally categorized into early gastric cancer and non-cancer groups depending on whether early gastric cancer lesions were present or had previously been identified. Early gastric cancer was defined based on endoscopic submucosal dissection (ESD) indications: (i) UL0 cT1a differentiated-type carcinomas; (ii) UL1 cT1a differentiated-type carcinomas with a long diameter ≤3 cm; or (iii) UL0 cT1a undifferentiated-type carcinomas with a long diameter ≤2 cm. Immunohistochemical staining was performed using an anti-H. pylori antibody (Beijing Zhongshan Golden Bridge Biotechnology Co., Ltd, Beijing, China). Positive results were graded as mild (1+): occasional bacteria or colonization in <1/3 of the specimen length; moderate (2+): colonization exceeding 1/3 but <2/3 of the specimen, or continuous but sparse distribution on the epithelial surface; and severe (3+): clusters of H. pylori distributed across the full length of the specimen. The gastric body and antrum were assessed separately, and distribution patterns were classified as gastric antrum > gastric body, gastric antrum = gastric body, or gastric body > gastric antrum. The distribution of H. pylori across subgroups was compared, and multivariate analyses were performed to identify risk factors associated with the development of early gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

* age 18-80 years
* received H. pylori immunohistochemical testing at our center and tested positive.

Exclusion Criteria:

* biopsies not collected from both the greater and lesser curvatures of the gastric antrum and body
* history of stomach surgery
* suspected autoimmune gastritis under endoscopy
* liver cirrhosis
* severe comorbidities such as advanced cancer or renal failure
* advanced gastric cancer or gastric lymphoma

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cases that underwent gastric H. pylori immunohistochemical staining at our center from March 1, 2023, to August 15, 2025.
Sampling Method: Non-Probability Sample
Enrollment: 231 (Estimated)
Dates: Start 2025-10-22 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The status of Helicobacter pylori(H. pylori) | one week after the endoscopic submucosal dissection (ESD)
  The status of H. pylori included negative and positive status. Positve results were graded as mild (1+): occasional bacteria or colonization in <1/3 of the specimen length; moderate (2+): colonization exceeding 1/3 but <2/3 of the specimen, or continuous but sparse distribution on the epithelial surface; and severe (3+): clusters of H. pylori distributed across the full length of the specimen. The gastric body and antrum were assessed separately.

SECONDARY OUTCOMES:
the percentage of H. pylori positive status of gastric antrum in early gastric cancer | one year after the endoscopic submucosal dissection (ESD)
  the percentage of H. pylori positive status of gastric antrum in early gastric cancer was assessed

OTHER OUTCOMES:
the percentage of H. pylori positive status of gastric body in early gastric cancer | one year after the endoscopic submucosal dissection (ESD)
  the percentage of H. pylori positive status of gastric body in early gastric cancer was assessed
the percentage of H. pylori positive status of gastric antrum in gastritis | one year after the endoscopic submucosal dissection (ESD)
  the percentage of H. pylori positive status of gastric antrum in gastritis was assessed
the percentage of H. pylori positive status of gastric body in gastritis | one year after the endoscopic submucosal dissection (ESD)
  the percentage of H. pylori positive status of gastric body in gastritis was assessed

CONTACTS AND LOCATIONS:
Locations (1):
- the First Hospital of Jilin University, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: No